CLINICAL TRIAL: NCT01169701
Title: Multicenter, Open-label, Randomized, 24 Months Follow-up, Two Arm Study to Compare the Efficacy of Everolimus in Improving the Cardiovascular Profile in a Regimen With Mycophenolic Acid vs. a Regimen of CNI+MPA in Maintenance Renal Transplant Recipients.
Brief Title: 24 Months Follow-up, Two Arm Study to Compare the Cardiovascular Profile in a Regimen With Everolimus + Mycophenolic Acid (MPA) Versus (vs.) a Regimen of CNI+MPA in Maintenance Renal Transplant Recipients
Acronym: EVITA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001AES07; 2009-013780-19 (EudraCT Number)
Record Dates: First submitted 2010-07-22; First posted 2010-07-26 (Estimated); Results first posted 2015-04-30 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-11

CONDITIONS: Renal Transplant
Keywords: Renal transplant, everolimus, cardiovascular profile, CNI-free immunosuppression, left ventricular hypertrophy, biopsy proved acute rejection (BPAR)
MeSH Terms: conditions — Hypertrophy, Left Ventricular | interventions — Everolimus; Tacrolimus; Mycophenolic Acid

ARMS (2):
- Tacrolimus (Active Comparator): Participants continued with the same tacrolimus+Mycophenolic acid (MPA) (Myfortic® or Cell-Cept®) doses that were taken before study initiation (tacrolimus levels 4-7 ng/ml).
  Interventions: Drug: Tacrolimus; Drug: Mycophenolic acid (MPA)
- Everolimus (Experimental): Participants received an initial dose (day 1) of Everolimus (EVL) 2mg at night and tacrolimus (if taking Prograf®, a full dose of Prograf® in the morning and a 50% dose of Prograf® at night; if taking Advagraf®, a 75% dose in the morning. On days 2 and 3, participants took EVL 2 mg twice daily (bid) without tacrolimus. On days 4 and 5, the EVL dose was adjusted and levels maintained between 5-8 ng/mL. Participants also continued with their MPA doses that were taken prior to study initiation.
  Interventions: Drug: Everolimus; Drug: Tacrolimus; Drug: Mycophenolic acid (MPA)

INTERVENTIONS:
Drug: Everolimus — Everolimus was supplied in boxes with 60 tablets. Available tablets: 1.0 mg, 0.5 mg and 0.25 mg.
  Other Names: Certican®
  Arms: Everolimus
Drug: Tacrolimus — Tacrolimus was administrated as Prograf® or Advagraf®, but could not be changed during study.
  Other Names: Prograf®, Advagraf®
Drug: Mycophenolic acid (MPA) — Myfortic® (MFS) was given as 720-1440 mg/day or 360-1440 mg/day. Cell-Cept® (MMF) was given as 1000-2000 mg/day or 500-2000 mg/day.
  Other Names: Myfortic®; Cell-Cept®

SUMMARY:
The objective of the study is to compare the cardiovascular profile of an everolimus and mycophenolic acid immunosuppressive regimen with a calcineurin inhibitor and mycophenolic acid regimen in maintenance renal transplant patients

ELIGIBILITY:
Inclusion Criteria:

* Received kidney transplant > 6 months and < 3 years prior to study enrollment
* Receiving immunosuppressive regimen that includes tacrolimus and mycophenolic acid
* Between 18 and 70 years of age
* Willing to provide written informed consent

Exclusion Criteria:

* Patients with an actual serum creatinine ≥ 2 mg/dl and/or eGFR≤ 40 ml/min and/or proteinuria≥ 500mg/day
* Patients who suffered from severe humoral and/or cellular rejection (≥ BANFF IIb, recurrent acute rejection or steroid resistant acute rejection in the previous years
* Patients who have severe hypercholesterolemia (>350 mg/dL; >9 mmol/L) or hypertriglyceridemia (>500 mg/dL; >8.5 mmol/L). Patients with controlled hyperlipidemia are acceptable.
* Diabetic patients
* Woman of child-bearing potential who is planning to become pregnant or is pregnant and/or lactating who is unwilling to use effective means of contraception
* Presence of psychiatric illness (i.e., schizophrenia, major depression) that, in the opinion of the site investigator, would interfere with study requirements
* Any other medical condition that, in the opinion of the site investigator based on recall or chart review would interfere with completing the study
* Receiving any investigational drug or have received any investigational drug within 30 days prior to study enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2010-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Spain (4):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid, Madrid

REFERENCES:
- [Derived] Cruzado JM, Pascual J, Sanchez-Fructuoso A, Seron D, Diaz JM, Rengel M, Oppenheimer F, Hernandez D, Paravisini A, Saval N, Morales JM; Evita Study Group. Controlled randomized study comparing the cardiovascular profile of everolimus with tacrolimus in renal transplantation. Transpl Int. 2016 Dec;29(12):1317-1328. doi: 10.1111/tri.12862. Epub 2016 Oct 17. PMID 27648523

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tacrolimus | Everolimus
Started | 36 | 35
Safety Set | 36 | 35
Intent to Treat (ITT) Set | 32 | 28
Completed | 31 | 25
Not Completed | 5 | 10
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Adverse Event | 1 | 2
Not completed — Exclusion criteria | 2 | 0
Not completed — Death | 0 | 1
Not completed — Administrative problems | 0 | 1
Not completed — Serious adverse event | 0 | 1
Not completed — Sponsor decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tacrolimus | Everolimus | Total
Number analyzed (Participants) | 36 | 35 | 71
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.1 (12.0) | 47.4 (13.2) | 48.3 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 29
  Male | 20 | 22 | 42

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Left Ventricular Mass Index (LVMI)
Description: Left ventricular hypertrophy grade was assessed by echocardiogram where the left ventricular mass index was calculated. The presence of LVM was defined as > 49.2 g/m^2.7 in men and >46.7 g/m^2.7 in women. A negative change from baseline indicates improvement.
Time Frame: Baseline, Month 24
Population: Participants from the Intent to Treat (ITT) analysis set, who had both baseline and month 24 values, were analyzed. The ITT included participants who received at least one dose of study medication and at least one post baseline LVMI value.
Measure: Mean (Standard Deviation); unit: g/m^2.7
Arm/Group | Tacrolimus | Everolimus
Number analyzed (Participants) | 31 | 25
g/m^2.7 | -6.071 (20.116) | -4.008 (17.610)

2. Secondary Outcome: Change From Baseline in Mean 24 Hour Systolic and Diastolic Blood Pressure
Description: Blood pressure was measured using ambulatory blood pressure monitoring (ABPM). A negative change from baseline indicates improvement.
Time Frame: Baseline, Month 6, month 12, month 24
Population: Participants from the safety analysis set were considered for this analysis. The safety analysis set included participants who received at least one dose of study medication. For each time point, only participants, who had values at both baseline and the given time point, were analyzed for that time point.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tacrolimus | Everolimus
Number analyzed (Participants) | 31 | 30
mmHg
  Month 6 (n=31,29) | -0.6 (9.1) | 3.2 (8.6)
  Month 12 (n=28,24) | 2.1 (6.9) | 2.7 (10.4)
  Month 24 (n=29,24) | 2.2 (10.6) | 2.0 (8.7)

3. Secondary Outcome: Pulse Wave Velocity (PWV)
Description: Utilizing the SphygmoCor Device, ECG leads placed at the carotid and femoral arteries provided the measure of the pulse wave at that particular arterial location. The distance between the two vascular beds divided by the pulse wave time shift provided a measure of the pulse wave velocity.
Time Frame: Month 6, month 24
Population: Participants from the safety analysis set were considered for this analysis. The safety analysis set included participants who received at least one dose of study medication. For each time point, only participants, who had values at the given time point, were analyzed for that time point.
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | Tacrolimus | Everolimus
Number analyzed (Participants) | 36 | 35
m/sec
  Month 6 (n=31,30) | 7.01 (1.62) | 7.40 (1.62)
  Month 24 (n=28,25) | 7.58 (1.68) | 7.06 (1.74)

4. Secondary Outcome: Percentage of Participants With Major Cardiovascular Events (MACE)
Description: The percentage of participants who experienced MACE were reported. MACE included acute myocardial infarction, insertion or replacement of implantable defibrillator, peripheral vascular disorders, congestive heart failure, coronary artery bypass, other events, percutaneous coronary intervention and stroke.
Time Frame: Month 24
Population: The Intent to Treat (ITT) analysis set: The ITT included participants who received at least one dose of study medication and had at least one post baseline LVMI value.
Measure: Number; unit: Percentage of participants
Arm/Group | Tacrolimus | Everolimus
Number analyzed (Participants) | 32 | 28
Percentage of participants | 0.00 | 0.00

5. Secondary Outcome: Renal Function Measured by Serum Creatinine
Description: Serum samples were collected to analyze serum creatinine.
Time Frame: Month 6, month 12, month 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Tacrolimus | Everolimus
Number analyzed (Participants) | 36 | 35
mg/dl
  Month 6 (n=33,29) | 1.232 (0.272) | 1.234 (0.360)
  Month 12 (n=32,28) | 1.231 (0.278) | 1.256 (0.367)
  Month 24 (n= 31,26) | 1.217 (0.235) | 1.260 (0.358)

6. Secondary Outcome: Renal Function as Measured by Creatinine Clearance
Description: Creatinine clearance was calculated using the Cockroft-Gault formula.
Time Frame: Month 6, month 12, month 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/min
Arm/Group | Tacrolimus | Everolimus
Number analyzed (Participants) | 36 | 35
mg/min
  Month 6 (n=29,25) | 64.841 (16.163) | 76.618 (27.708)
  Month 12 (n=28,25) | 65.037 (15.866) | 73.363 (25.989)
  Month 24 (n=28,24) | 66.933 (13.264) | 72.910 (23.926)

7. Secondary Outcome: Renal Function as Measured by Estimated Glomerular Filtration Rate (eGFR)
Description: Estimated GFR was caluclated using the modification of diet in renal disease (MDRD) formula.
Time Frame: Month 6, month 12, month 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Tacrolimus | Everolimus
Number analyzed (Participants) | 36 | 35
mL/min/1.73m^2
  Month 6 (n=33,29) | 55.648 (11.244) | 63.781 (18.380)
  Month 12 (n=32,28) | 57.757 (11.391) | 61.225 (19.239)
  Month 24 (n=31,26) | 57.727 (10.498) | 60.779 (17.023)

8. Secondary Outcome: Change From Baseline in Cardiovascular Biomarkers: Troponin I and Collagen Type 1 C-telopeptide (ICTP)
Description: Blood samples were collected to analyze Troponin I and collagen type 1 C-telopeptide (ICTP). A negative change from baseline indicates improvement.
Time Frame: Baseline, month 6, month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Tacrolimus | Everolimus
Number analyzed (Participants) | 36 | 35
ng/ml
  Troponin 1, Month 6 (n=27,30) | 0.000 (0.010) | -0.006 (0.026)
  Troponin 1, Month 24 (n=24,24) | 0.003 (0.026) | -0.007 (0.018)
  ICTP, Month 6 (n=27,30) | 0.049 (0.341) | -0.195 (0.234)
  ICTP, Month 24 (n=24,24) | -0.035 (0.366) | -0.125 (0.323)

9. Secondary Outcome: Change From Baseline in the Cardiovascular Biomarker, Glycosylated Hemoglobin (HbA1c)
Description: Blood samples were collected to analyze HbA1c. A negative change from baseline indicates improvement.
Time Frame: Baseline, month 6, month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Tacrolimus | Everolimus
Number analyzed (Participants) | 36 | 35
Percentage of HbA1c
  Month 6 (n=20,22) | 0.015 (0.184) | 0.159 (0.346)
  Month12 (n=22,20) | 0.045 (0.237) | 0.185 (0.407)

10. Secondary Outcome: Change From Baseline in the Cardiovascular Biomarker, Myeloperoxidase (MPO)
Description: Blood samples were collected to analyze MPO. A negative change from baseline indicates improvement.
Time Frame: Baseline, month 6, month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Tacrolimus | Everolimus
Number analyzed (Participants) | 36 | 35
U/mL
  Month 6 (n=27,30) | 0.433 (2.189) | -0.093 (1.158)
  Month 24 (n=24,24) | -0.329 (0.280) | -0.642 (0.972)

11. Secondary Outcome: Change From Baseline in the Cardiovascular Biomarker, N-terminal Pro-brain Natriuretic Peptide Fraction (NT-proBNP)
Description: Blood samples were collected to analyze NT-proBNP. A negative change from baseline indicates improvement.
Time Frame: Baseline, month 6, month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tacrolimus | Everolimus
Number analyzed (Participants) | 36 | 35
pg/mL
  Month 6 (n=27,30) | 21.604 (294.82) | -79.10 (401.44)
  Month 24 (n=24,24) | -80.20 (424.24) | -193.3 (590.90)

12. Secondary Outcome: Change From Baseline in the Cardiovascular Biomarker, Type 1 Procollagen Amino-terminal-propeptide (PINP)
Description: Blood samples were collected to analyze PCR. A negative change from baseline indicates improvement.
Time Frame: Baseline, month 6, month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/l
Arm/Group | Tacrolimus | Everolimus
Number analyzed (Participants) | 36 | 35
ug/l
  Month 6 (n=27,30) | -13.82 (34.110) | -33.36 (33.227)
  Month 24 (n=24,24) | -13.65 (40.675) | -28.17 (30.381)

13. Secondary Outcome: Change From Baseline in Cardiovascular Biomarkers, C-reactive Protein (CRP)
Description: Blood samples were collected to analyze CRP. A negative change from baseline indicates improvement.
Time Frame: Baseline, month 6, month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Tacrolimus | Everolimus
Number analyzed (Participants) | 36 | 35
mg/dl
  Month 6 (n=27,30) | 0.512 (2.342) | 0.326 (1.129)
  Month 24 (n=24,24) | 0.100 (0.469) | -0.040 (1.683)

14. Secondary Outcome: Percentage of Participants With Biopsy-proven Acute Rejection (BPAR), Graft Loss, Death and Lost to Follow up
Description: The incidence of BPAR, graft loss, death and lost to follow-up events was calculated using relative frequency.
Time Frame: Month 24
Population: Intent to Treat (ITT): The ITT included participants who received at least one dose of study medication and at least one post baseline LVMI value.
Measure: Number; unit: Percentage of participants
Arm/Group | Tacrolimus | Everolimus
Number analyzed (Participants) | 32 | 28
Percentage of participants
  BPAR | 0.00 | 0.00
  Graft loss | 0.00 | 0.00
  Deaths | 0.00 | 0.00
  Lost to follow-up | 3.13 | 0.00

ADVERSE EVENTS:
Arm/Group | Tacrolimus | Everolimus
Serious Adverse Events (participants affected / at risk) | 5/36 | 8/35
Other Adverse Events (participants affected / at risk) | 21/36 | 24/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus (N=36) | Everolimus (N=35)
Pyrexia (General disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Arteriovenous fistula operation (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus (N=36) | Everolimus (N=35)
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 2
Polycythaemia (Blood and lymphatic system disorders) | 1 | 2
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 4 | 3
Asthenia (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 3 | 6
Bronchitis (Infections and infestations) | 2 | 0
Escherichia urinary tract infection (Infections and infestations) | 4 | 4
Nasopharyngitis (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 0 | 2
Respiratory tract infection (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 7 | 1
Urinary tract infection bacterial (Infections and infestations) | 1 | 2
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 0
Dizziness (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 2 | 2
Depression (Psychiatric disorders) | 0 | 2
Proteinuria (Renal and urinary disorders) | 0 | 5
Metrorrhagia (Reproductive system and breast disorders) | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.